CLINICAL TRIAL: NCT02126410
Title: Associations Between Self-Reported Sleep Duration and Sarcopenia in Community-Dwelling Older Adults
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201402038RINB
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Community-Based Participatory Research; Aged; Sleep; Body Composition
Keywords: sarcopenia; sleep duration; body composition; skeletal muscle
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1. BACKGROUNDS: Currently, elderly people comprise more than 10% of the total Taiwanese population. However, within the context of self-reported sleep duration and health risks, research into the association between sleep duration and body composition changes in older people is limited. It is important to gain an understanding of such an association of older people to estimate the public health burden.
2. OBJECTIVES: To assess the association between self-reported sleep duration and sarcopenia as well as obesity in community-dwelling older adults.
3. HYPOTHESIS: Self-reported sleep duration is associated with prevalence of sarcopenia and obesity in community-dwelling older adults.
4. DESIGN: A cross-sectional investigation.
5. SETTING: Communities in Zhongzheng district, Taipei.
6. PARTICIPANTS: Four hundred and forty-eight community-dwelling adults (224 men and 264 women) aged 65 years and older.
7. MEASUREMENTS: The investigators evaluated self-reported sleep duration by deriving from the Pittsburgh Sleep Quality Index and 7-d recall physical activity diary. Skeletal muscle mass was estimated by the predicted equation from a bioelectrical impedance analysis measurement. The Groningen Activity Restriction Scale and the Chinese Geriatric Depression Screening Scale were used to evaluate physical disability and depression, respectively.

ELIGIBILITY:
1. hyper- or hypothyroidism.
2. taking prescribed medications (such as growth hormone, testosterone, or progesterone) known to alter body composition.
3. any condition that prevented them from completing our questionnaires or the functional capacity test (e.g., amputee, nonambulatory even with the use of a walker or a cane, blind, or deaf).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: community-dwelling elderly (>= 65 years old)
Sampling Method: Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass index | one day
  Using Bioelectrical Impedance Analysis to measure skeletal muscle mass (kg) and further calculate skeletal muscle mass index to investigate the prevalence of sarcopenia.

SECONDARY OUTCOMES:
Sleep quality | one day
  Using Pittsburgh Sleep Quality Index to record the sleep quality
Level of physical activity | one day
  Using 7-d recall physical activity questionnaire to evaluate general physical activity in the past 7 days.
Sleep duration | one day
  Recording the sleep time at night and daytime napping separately.
Body composition | one day
  Using Bioelectrical Impedance Analysis to measure fat percentage in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, Ph.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan, Taiwan